CLINICAL TRIAL: NCT04806984
Title: Improving Gap Closure Rates Using a Predictive Model
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-CIN Gaps Predictive Model
Record Dates: First submitted 2021-03-05; First posted 2021-03-19 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Communication; Appointments and Schedules
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Call center phone call: Participants randomized to this arm will receive a phone call from the call center reminding them to schedule their appointments.
  Interventions: Other: Participant outreach
- No call center phone call: Participants randomized to this arm will not receive a phone call from the call center reminding them to schedule their appointments.
- MyChart message: Participants randomized to this arm will receive an automated MyChart message reminding them to schedule their appointments.
  Interventions: Other: Participant outreach
- No MyChart message: Participants randomized to this arm will not receive an automated MyChart message reminding them to schedule their appointments.

INTERVENTIONS:
Other: Participant outreach — Participants in the experimental arms will receive a call center phone call or MyChart message to remind them to schedule their appointments.
  Groups: Call center phone call; MyChart message

SUMMARY:
NYU Langone Health outreaches to patients to remind them to schedule their appointments by phone or MyChart message.The proposed study will test different outreach methods using a predictive risk model. The goal is to increase gap closure rate by the end of the year.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the NYU Langone network who are due for gaps in care.

Exclusion Criteria:

* Patients in the NYU Langone network are not due for gaps in care.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the NYU Langone network
Sampling Method: Non-Probability Sample
Enrollment: 34896 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Gap closure rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No